CLINICAL TRIAL: NCT03806530
Title: DIalysis Symptom COntrol-Restless Legs Syndrome Trial (DISCO-RLS Trial): A Randomized Controlled Trial
Brief Title: DIalysis Symptom COntrol-Restless Legs Syndrome Trial
Acronym: DISCO-RLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DISCO_RLS_001
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: End Stage Renal Disease; Restless Legs Syndrome
MeSH Terms: conditions — Kidney Failure, Chronic; Restless Legs Syndrome | interventions — Gabapentin; ropinirole

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to 1 of 8 treatment sequences. Each sequence is composed of 4 periods and in each period participants will receive 1 of 4 possible combinations of study medications (gabapentin+ropinirole, gabapentin+placebo ropinirole, ropinirole+placebo gabapentin, placebo gabapentin+placebo ropinirole).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study interventions will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gabapentin + Ropinirole (Active Comparator): Gabapentin 100 mg capsule, once daily for 4 weeks. Ropinirole 0.50 mg capsule, once daily for 4 weeks.
  Interventions: Drug: Gabapentin; Drug: Ropinirole
- Gabapentin + Placebo Ropinirole (Placebo Comparator): Gabapentin 100 mg capsule, once daily for 4 weeks. Ropinirole placebo 0.50 mg capsule, once daily for 4 weeks.
  Interventions: Drug: Gabapentin; Drug: Placebo Ropinirole
- Ropinirole + Placebo Gabapentin (Placebo Comparator): Gabapentin placebo 100 mg capsule, once daily for 4 weeks. Ropinirole 0.50 mg capsule, once daily for 4 weeks.
  Interventions: Drug: Ropinirole; Drug: Placebo Gabapentin
- Placebo Gabapentin + Placebo Ropinirole (Placebo Comparator): Gabapentin placebo 100 mg capsule, once daily for 4 weeks. Ropinirole placebo 0.50 mg capsule, once daily for 4 weeks.
  Interventions: Drug: Placebo Gabapentin; Drug: Placebo Ropinirole

INTERVENTIONS:
Drug: Gabapentin — 100 mg capsule
  Other Names: GD-Gabapentin
  Arms: Gabapentin + Placebo Ropinirole; Gabapentin + Ropinirole
Drug: Ropinirole — 0.50 mg capsule
  Other Names: pms-Ropinirole
  Arms: Gabapentin + Ropinirole; Ropinirole + Placebo Gabapentin
Drug: Placebo Gabapentin — Placebo capsule
  Other Names: Placebo
  Arms: Placebo Gabapentin + Placebo Ropinirole; Ropinirole + Placebo Gabapentin
Drug: Placebo Ropinirole — Placebo capsule
  Other Names: Placebo
  Arms: Gabapentin + Placebo Ropinirole; Placebo Gabapentin + Placebo Ropinirole

SUMMARY:
The DISCO-RLS Trial is a randomized controlled trial to determine the safety and efficacy of pharmacologic therapy (ropinirole versus placebo and gabapentin versus placebo) for the treatment of Restless Legs Syndrome in patients with End Stage Renal Disease requiring hemodialysis.

DETAILED DESCRIPTION:
The DISCO-RLS Trial is a randomized controlled trial to determine whether or not a fixed, low-dose therapy with ropinirole and/or gabapentin is safe and effective compared to either alone or placebo for the treatment of Restless Legs Syndrome in patients with End Stage Renal Disease receiving hemodialysis. DISCO-RLS will randomize a total of 80 participants. Participants will be randomized to 1 of 8 treatment sequences. Each sequence is composed of 4 periods and in each period participants will receive 1 of 4 possible combinations of study medications (gabapentin+ropinirole, gabapentin+placebo ropinirole, ropinirole+placebo gabapentin, placebo gabapentin+placebo ropinirole). Eligible participants will complete a 1-week Run-In period followed by 4 periods of 4 weeks each for a total of 16-week follow-up after randomization. A final study visit will be completed at the end of the 16 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years
* Has received at least 90 days of in-center hemodialysis at a frequency at least 3 times weekly
* RLS defined by 2012 Revised International Restless Legs Syndrome Study Group (IRLSSG) Diagnostic Criteria for RLS and of moderate severity defined by an IRLS score greater or equal to 10 with symptoms more than 2 days per week (see IRLS question #7)
* Provides informed consent

Exclusion Criteria:

* Hemoglobin<80g/L in the previous 4 weeks
* Intolerance to a dopamine agonists (e.g. pramipexole or ropinirole) or alpha 2 delta ligands (e.g. gabapentin, Neurontin, pregabalin, or Lyrica)
* Change in medication to treat RLS in previous 4 weeks
* Current pregnancy
* Planned kidney transplantation, travel or relocation in the next 6 months
* Unable to complete RLS symptom and HRQOL measurements due to language barrier or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group Rating Scale (IRLS) | 18 weeks (Baseline, Run-In, Follow-up)
  The IRLS is a measure of severity of Restless Legs Syndrome. It includes 10 items, measured on a scale of 0-4. A score of 1-10 indicates mild severity, 11-20 indicates moderate severity, 21-30 is severe and 31-40 is very severe. Primary outcome is the difference in IRLS scores for each of the treatment regimens.

SECONDARY OUTCOMES:
Restless Legs Syndrome-6 Scale (RLS-6) | 18 weeks (Baseline, Run-In, Follow-up)
  The RLS-6 is a measure of severity of Restless Legs Syndrome for the past week. It includes 6 items, measured on a scale of 0-10. Each item is measured from no symptoms (score of 0) to very severe symptoms (score of 10). Secondary outcome is the difference in RLS-6 scores for each of the treatment regimens.
Patient Global Impressions (PGI) | 18 weeks (Baseline, Run-In, Follow-up)
  The PGI is a measure of Restless Legs Syndrome symptom severity. It includes 1 item, measured on a scale of 1-7. 1 indicates mild severity, 3 indicates moderate severity, 5 is severe and 7 is very severe. Secondary outcome is the difference in PGI scores for each of the treatment regimens
Euro-Quality of Life Scale (EQ-5D-5L) | 18 weeks (Baseline, Run-In, Follow-up)
  The EQ-5D-5L is a measure of health status. It includes 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and a visual analogue scale of 0-100 (0 being worst health and 100 being best health). The scale is measured by levels. Level 1 indicating no problems, 2 indicating slight problems, 3 indicating moderate problems, 4 indicating severe problems and 5 indicating extreme problems. Secondary outcome is the difference in EQ-5D-5L scores for each of the treatment regimens
Incidence of falls, fractures and hospitalizations/emergency room visits due to altered level of consciousness. | 18 weeks (Baseline, Run-In, Follow-up)
  The total number of falls, fractures, or hospitalization/emergency rooms visits due to confusion/delirium or altered mental state.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Walsh, PhD,FRCPC(C), Principal Investigator — Population Health Research Institute, McMaster University
Locations (3):
- Canada (3):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - St. Joseph's Hamilton Healthcare, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collister D, Pohl K, Herrington G, Lee SF, Rabbat C, Tennankore K, Zimmermann D, Tangri N, Wald R, Manns B, Suri RS, Nadeau-Fredette AC, Goupil R, Silver SA, Walsh M. The DIalysis Symptom COntrol-Restless Legs Syndrome (DISCO-RLS) Trial: A Protocol for a Randomized, Crossover, Placebo-Controlled Blinded Trial. Can J Kidney Health Dis. 2020 Nov 26;7:2054358120968959. doi: 10.1177/2054358120968959. eCollection 2020. PMID 33294203